CLINICAL TRIAL: NCT05555342
Title: A Novel Method for Treating Lung Metastases With the Combination of Electrical Fields and Radiation Therapy: A Single-Arm Pilot Study
Brief Title: A Novel Method for Treating Lung Met w/Combo of Electric Fields & Rad Therapy: A Single-Arm
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Jeremy Harris, Assistant Professor of Clinical Radiation Oncology, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1723; UCI 21-222 (Other: CFCCC)
Record Dates: First submitted 2022-09-20; First posted 2022-09-26 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Lung Tumor; Metastatic Cancer
Keywords: lung metastasis; Stereotactic Ablative Radiotherapy; Percutaneous ablation; irreversible electroporation
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis | interventions — Electroporation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- IRE ablation and radiation therapy (Experimental): Patients will be treated with IRE ablation directed at the target lesion on day 1. Moderate-dose, single-fraction radiation therapy will be delivered to the target lesion on day 8 to day 15.
  Interventions: Procedure: Irreversible electroporation (IRE) ablation; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Irreversible electroporation (IRE) ablation — IRE will be performed using the NanoKnife or Aliya System. CT or cone-beam CT will be used to direct electrode placement.
Radiation: Radiation Therapy — Moderate-dose radiation therapy to the target tumor(s) in 1 fraction.

SUMMARY:
This is a phase 0, pilot prospective study to determine the feasibility of combined irreversible electroporation (IRE) and radiation therapy in subjects with lung tumors with metastatic cancer of any histology. These are subjects who have advanced disease (stage IV) or previously treated disease that has become progressive, recurrent, or metastatic.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic cancer of any histology. There must be a lung tumor present, although the lung tumor does not specifically need to have been biopsied.
* Patients must have advanced disease (stage IV) or previously treated disease that has become progressive, recurrent, or metastatic.
* Patients may have received any number of prior systemic or local therapies. There will be no prespecified washout period prior to IRE. However, systemic therapy will be halted while receiving IRE and radiation, and can be restarted following completion of radiation therapy.
* Up to 3 lesions may be included for treatment. The selected lesion(s) should be amenable to ablation and irradiation and patients will be eligible for ablation and irradiation in the judgment of the treating radiologist and radiation oncologist. If more than one lesion is selected, they should be separated by at least 5 cm to minimize lung irradiation. The target lesion for treatment by IRE and radiation will be a tumor not previously treated by radiation. This target lesion must be measurable, defined as the ability to be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >10 mm with spiral CT scan. The upper limit to the target lesion is 6 cm maximal diameter, but it also must be planned to be encompassed entirely by an IRE ablative zone. Any number of IRE probes will be allowed such that the entire tumor can be ablated.
* Must be age ≥ 18 years. Children are excluded from this study but will be eligible for future pediatric trials, if applicable.

  1. Both men and women and members of all races and ethnic groups are eligible for this trial. Non-English speaking, deaf, hard of hearing and illiterate individuals are eligible for this trial.
* Performance status: ECOG performance status ≤2 (Karnofsky ≥50%).
* Life expectancy of ≥3 months.
* Adequate organ and marrow function as defined below. Labs should be performed within 14 days of treatment.

  1. Platelets ≥50,000/mcL
  2. Hemoglobin ≥8 g/dL
  3. Absolute neutrophil count ≥1,000/mcL
  4. INR <1.5
* Female patients of childbearing potential must have a negative urine or serum pregnancy during screening. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* The effects of ionizing radiation (i.e. radiation therapy) on the developing human fetus are known to have the potential for congenital abnormalities and fetal harm. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and until completion of radiation therapy. Should a woman become pregnant or suspect she is pregnant during this period, she should inform her treating physician immediately.

  1. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
  1. Has not undergone a hysterectomy or bilateral oophorectomy; or
  2. Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Patients must not have a history of (non-infectious) pneumonitis that required steroids or have current pneumonitis.
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Patient's whose target lesion has been previously treated with radiation therapy.
* Patients who have not recovered from adverse events due to prior anti-cancer therapy administered.
* Patients may not be receiving any other investigational agents 2 weeks prior to enrollment and until end of all therapeutic interventions.
* Patients with cardiac arrhythmias, pacemakers, or implanted defibrillator.
* Patients with epilepsy.
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients must not be pregnant due to the potential for congenital abnormalities and fetal harm caused by ionizing radiation.
* Patients with disease amenable to curative intent therapy.
* Patient has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2024-10-27 (Actual)

PRIMARY OUTCOMES:
Feasibility, measured as the number of patients completing both IRE and the single fraction of radiation | Up to 3 years
  Number of patients completing treatment of both IRE and the single fraction of radiation. Up to 6 replacements are allowed (total subjects 6-12)

SECONDARY OUTCOMES:
Number of grade 3-5 adverse events | Up to 3 years
  Severe toxicity will be measured by cumulative CTCAE v5.0 grade 3-5 events. Evaluation of Grade 3-5 toxicity will be made at 30 days
Local failure at the treated site | Up to 3 years
  Local failure rate at the treated site will be determined using cumulative incidence rates with death as a competing event at 12 months after initiation of treatment
Duration of response | Up to 3 years
  The duration of response is measured from the time of treatment initiation until local failure is objectively documented
Progression-free survival | Up to 3 years
  Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Estimates at 6 and 12 months will be made.
Overall survival | Up to 3 years
  The duration of time from start of treatment to time of progression or death, whichever occurs first. Estimates at 6 and 12 months will be made.
Number of grade 1-5 adverse events | Up to 3 years
  Toxicity will be measured by cumulative CTCAE v5.0 grade 1-5 events. Evaluation of Grade 1-5 toxicity will be made at 30 days
Patient reported quality of life | Up to 3 years
  Mean summary score of the Functional Assessment of Cancer Therapy-Lung (FACT-L). Functional Assessment of Cancer Therapy-Lung (FACT-L) Scale is a 36-item self-reported instrument that measures multidimensional quality of life for lung cancer patients. Questions are scored on a 5-point Likert Scale. The FACT-L includes the FACT-G (general) assessment which is comprised of four subscales including Physical Well-Being (score = 0-28), Social/Family Well-Being (score= 0-28), Emotional Well Being (score = 0-24), and Functional Well-Being (score = 0-28), for a total score min/max = 0-108, plus, the Lung Cancer Subscale (nine lung cancer related items, score = 0-45). Total scores range from 0-136, with higher scores indicating better quality of life.
Forced vital capacity | Up to 3 years
  Pulmonary function is assessed by the volume change (mL) in the value of forced vital capacity (FVC)
Forced expiratory volume at 1 second (FEV1) | Up to 3 years
  Pulmonary function is assessed by volume change (mL) in the value of forced expiratory volume at 1 second (FEV1)
Diffusing capacity for carbon monoxide (DLCO) | Up to 3 years
  Pulmonary function is assessed by change in the value of diffusing capacity for carbon monoxide (DLCO) measured in mL/min/kPa

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Harris, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center University of California, Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harris JP, Boyd C, Shi M, Reilly M, Simon A, Seyedin SN, Chen WP, Nagasaka M, Nabar R, Abi-Jaoudeh N. Pilot Study of Combining Stereotactic Body Radiation Therapy with Pulsed Field Ablation for Oligometastatic/Oligoprogressive Lung Tumors. J Vasc Interv Radiol. 2025 Nov;36(11):1687-1695. doi: 10.1016/j.jvir.2025.08.005. Epub 2025 Aug 11. PMID 40803526